CLINICAL TRIAL: NCT00555230
Title: Effects of HMG-coA Reductase Inhibitor on Progression of Carotid Intima-Media Thickness and Arterial Stiffness in Rheumatoid Arthritis
Brief Title: Effects of HMG-coA Reductase Inhibitor on Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Edumun K Li,MD, the Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-2007-004
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
Keywords: HMG-CoA reductase inhibitors; Crestor; Rosuvastatin
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 5mg daily for 4 weeks then step up to 10mg or matching placebo for 52 weeks
  Other Names: crestor
  Arms: 1
Drug: Placebo — 5mg daily for 4 weeks then step up to 10mg or matching placebo for 52 weeks
  Other Names: crestor
  Arms: 2

SUMMARY:
The purpose of this study is:

1. To evaluate the prevalence of preclinical atherosclerosis in Chinese patients with RA compared to healthy controls.
2. To determine those clinical and biological measures that best predict the presence of plaque and increased arterial stiffness.
3. To ascertain the efficacy and safety of rosuvastatin in the prevention of atherosclerosis in patients with RA measured by carotid intima-media thickness (IMT) and pulse wave velocity (PWV).

DETAILED DESCRIPTION:
150 consecutive RA patients followed at the Rheumatology clinic of the Prince of Wales Hospital will be recruited for this double-blind, randomized, placebo-control trial. Patients were matched to 150 controls on the basis of age (within 5 years), sex, body mass index (+/-5Kg) and ethnicity for the cross sectional study on the prevalence of subclinical atherosclerosis. Controls were healthy individuals recruited from the same community who underwent similar imaging protocols of the IMT and PWV assessments.

Primary outcome is the improvement of atherosclerosis by Rosuvastatin therapy, evaluated by IMT and PWV.

Secondary outcomes:

* Prevalence of premature atherosclerosis in RA patients compared to healthy controls in terms of the presence of plague and PWV.
* Correlation between clinical parameters, inflammatory markers (CRP/hsCRP, TNF-alpha and IL-6) and atherosclerosis (evaluated by IMT, the presence of plaque and PWV).
* Relation among PWV, ABI and AI in RA patients, and clinical significance of their combination.
* Determine which segment's PWV has a better relation with RA disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 years of age or older
* Clinical diagnosis of RA with a duration of at least 6 month
* Prednisolone < =10 mg/day
* NSAID or DMARD
* Informed consent

Exclusion Criteria:

* Little or no ability for self-care
* Type 1 diabetes mellitus
* Uncontrolled hypertension(> 160/95 mmHg)
* Total cholesterol > 240 mg/dl, current or recent (within the past 3 months)
* History of coronary bypass grafting, myocardial infraction within 28days, left ventricular dysfunction (ejection fraction < 40%), significant valvular heart disease
* Current treatment with ACE inhibitor, angiotensin II receptor blockers or beta-blockers, lipid lowering drug, or contra-indication to statins
* Current treatment of oral contraceptives, estrogen and progestin was allowed but patient not willing to stop during study
* Current treatment with antioxidant therapy (Vitamin C or multivitamin)
* Received intra-articular, intramuscular, or intravenous corticosteroids in the past 4 weeks before screening
* Clinically significant renal disease(serum creatinine level ≥ 270 µmol/L) or aspartate aminotransferase(AST), alanine aminotransferase ALT), or creatine kinase (CK)≥ 2 X ULN
* Female of childbearing potential, unwilling to use adequate contraception during the study
* Current or recent (within the past 3 months) pregnancy and cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Improvement of atherosclerosis by Rosuvastatin therapy, evaluated by IMT and PWV. | baseline,week24,week52

SECONDARY OUTCOMES:
physical examination,blood pressure,pulse rate,and body weight measurements at each visit.Liver function and CK are performed at baseline,week 12,24 and 52.Correlation between clinical parameters,inflammatory markers and atherosclerosis. | baseline,week0,week3,week8,week12,week24,week36,week52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Kwok Ming Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- School of Pharmacy CUHK, Hong Kong, China